CLINICAL TRIAL: NCT05947968
Title: Scapular Proprioception Neuromuscular Facilitation Versus Shoulder Strengthening Exercises in Patients With Lateral Epicondylitis.
Brief Title: Scapular PNF Versus Shoulder Strengthening Exercises in Patients With Lateral Epicondylitis.
Acronym: PNF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahmoud Essam Abu Elfetouh Ghallab (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Mahmoud Essam Abu Elfetouh Ghallab, researcher, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Lateral epicondylitis
Record Dates: First submitted 2023-07-09; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Lateral Epicondylitis
Keywords: scapular PNF; scapular proprioceptive neuromuscular facilitation exercise; shoulder strengthening exercises
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Scapular PNF) (Experimental): will receive scapular proprioceptive neuromuscular facilitation exercise plus conventional treatment of lateral epicondylitis for 12 sessions (3 sessions per week for four weeks).
  The conventional treatment of lateral epicondylitis will be:
  1. Pulsed ultrasound over the lateral epicondyle for 5 min.
  2. Five minutes of deep friction massage. It will be consisted of deep circular motions using the fingertips over the area of maximal tenderness at the lateral epicondyle.
  3. Stretching exercise for extensor carpi radialis longus and brevis for 3 repetitions, each repetition will be 45 seconds with 30 seconds' rest.
  4. Strengthening exercise for wrist extensors, eccentric exercise for wrist extensors will be as follow: 3 sets, 10 repetitions, 1 min rest interval between each set.
  Interventions: Other: Scapular PNF
- Group B (Shoulder exercises) (Experimental): will receive shoulder strengthening exercise plus conventional treatment of lateral epicondylitis for 12 sessions (3 sessions per week for four weeks).
  Same conventional treatment in group (A)
  Interventions: Other: Shoulder strengthening exercises

INTERVENTIONS:
Other: Scapular PNF — Scapular proprioceptive neuromuscular facilitation exercise: will be applied in two diagonals:
  1. anterior elevation and posterior depression
  2. posterior elevation and anterior depression for 3 sets of 10 repetitions, The rest interval between sets will be 20 seconds.
  Patients will lay on the unaffected side while the therapist stands in the line of desired motion. Firstly, the therapist will give preparatory instructions. In the beginning of the pattern, the therapist pulls the scapula to the elongated position and then gives instructions for the desired movement.
  Arms: Group A (Scapular PNF)
Other: Shoulder strengthening exercises — Shoulder strengthening exercises:
  The following four exercises will focus on shoulder and scapular strengthening. Before starting the program, the patients will be thoroughly instructed in the four exercises, and illustrations with specific exercise instructions will be provided. All subjects will perform the exercises with the affected side for three sets of 10 repetitions for each exercise, with a 1-minute rest between sets.
  1. Standing shoulder external rotation with elastic resistance.
  2. Bilateral external rotation with scapular retraction exercise.
  3. Resisted scapular retraction with shoulder external rotation (Middle trapezius muscle).
  4. Weighted scapular retraction and downward rotation Y-shape (lower trapezius muscle).
  Arms: Group B (Shoulder exercises)

SUMMARY:
The purpose of this study is to compare between the effect of scapular proprioceptive neuromuscular facilitation versus shoulder and scapular strengthening exercise on pain, functional outcome and grip strength in patients with lateral epicondylitis.

DETAILED DESCRIPTION:
There is no standard treatment for lateral epicondylitis, it is always a combination of physical therapy modalities aimed to reduce pain and increase the ability to return functional activities participation. Accordingly, many researchers have added shoulder strengthening exercise to the rehabilitation plan for treating lateral epicondylitis.

Consequently, development of new concept of scapula motor control exercise using proprioceptive neuromuscular facilitation to add proximal stability to patients with lateral epicondylitis may be beneficial. We believe that this study can serve as a step toward documenting the evidence of scapular proprioceptive neuromuscular facilitation exercise in the treatment of patients with lateral epicondylitis which was not available before.

Patients with lateral epicondylitis will be recruited after approval of ethical committee of the faculty of physical therapy, Cairo University. All participants will sign a written informed consent form. After group assignment, patients' demographics will be collected, and then assessment of pain, function and grip strength will be performed. The same assessment procedure will be conducted by the end of the treatment (by the end of the 12th visit).

The study will be two comparative groups, pre-post experimental design, the subjects will be randomly assigned into one of two groups:

* Group (I) : will receive scapular proprioceptive neuromuscular facilitation exercises.
* Group (II) : will receive shoulder strengthening exercises.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included if they have the following criteria:

  * Fifty-two male and female subjects.
  * Patients complaining of chronic lateral epicondylitis (more than three months).
  * Age between 20-50.

Exclusion Criteria:

* Patients will be excluded if they had any of the following conditions:

  * Received physiotherapy in last 3 months.
  * Received corticosteroids injection in lateral epicondyle in last 3 months.
  * Receiving anti-inflammatories medications on regular basis.
  * Had neurologic problems in shoulder, neck and thoracic regions.
  * Had history of rheumatic disease.
  * Had cooperation difficulties due to cognitive disorders. All Patients will be instructed to keep away from activities that aggravate the symptoms such as grasping, lifting, knitting and using a screwdriver during the treatment period.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Pain intensity by The Numeric Pain Rating Scale (NPRS) | one month
  (NPRS) is a unidimensional measure of pain intensity in adults. Consists of 11-item NPRS. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g., "no pain") to '10' representing the other pain extreme (e.g., "pain as bad as you can imagine" or "worst pain imaginable.
Pain and functional disability by patient-rated tennis elbow evaluation (PRTEE) | one month
  The PRTEE is a valid and reliable tool that may be used in both research and clinical settings to assess the subjective outcome in patient with lateral epicondylitis. Subjects will be asked to rate the level of discomfort and difficulty they had encountered in the previous week. High total scores imply more pain and impairment; the scale spans from 0 to 100.
  The PRTEE is a 15-item questionnaire designed to measure forearm pain and disability in patients with LE. The PRTEE allows patients to rate their levels of pain and disability from 0 to 10, and consists of 2 subscales:
  1. PAIN subscale (0 = no pain, 10 = worst imaginable)
     • Pain - 5 items
  2. FUNCTION subscale (0 = no difficulty, 10 = unable to do)
     * Specific activities - 6 items
     * Usual activities - 4 items
Grip strength by Jammar handheld dynamometer. | one month
  The Jammar hand grip dynamometer is valid and reliable, will be used to assess the subject's pain-free grip strength while they are lying on their side with their elbow extended and pronated. Subjects will be instructed to squeeze the dynamometer handles until they experienced pain. It will be performed three times with 20 s rest period between repetitions. Average of three trials will be recorded in kilograms.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided